CLINICAL TRIAL: NCT02758158
Title: Clinical Evaluation of a Prototype Tri-modal Imaging Instrument for Thyroid Cancer
Brief Title: Tri-modal Imaging Instrument for Thyroid Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-9101
Record Dates: First submitted 2016-03-09; First posted 2016-05-02 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Thyroid Neoplasms; Thyroid Cancer; Thyroid Nodule
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tri-modal imaging (Experimental): Ultrasound and photoacoustic imaging of thyroid and adjacent lymph nodes. Imaging time: Approximately 30 minutes
  Interventions: Device: Tri-modal imaging

INTERVENTIONS:
Device: Tri-modal imaging — This trimodal imaging system was developed in collaboration with Sogang University and is composed of three subsystems: ultrasound, photoacoustic and fluorescence. For this study, the fluorescence subsystem will not be used. The photoacoustic and ultrasound subsystems and data acquisition are controlled by a single workstation. The complete system is Canadian Standards Association (CSA) certified.

SUMMARY:
Thyroid cancer affects 6,000 Canadians each year. Nodules on the thyroid are detected using ultrasound imaging and surgery is the most common treatment. However, most nodules are benign, and therefore a biopsy is needed to decide whether surgery is necessary. Ultrasound imaging is very sensitive for localizing nodules, but does not differentiate between cancerous and benign ones. To address this limitation of US imaging, investigators have designed and constructed, in collaboration with Sogang University, Seoul, S. Korea, a novel imaging system that performs complimentary imaging modalities (ultrasound (US), photoacoustic (PA)) that could potentially help diagnose nodules without the need for biopsy and unnecessary surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with thyroid nodules (cancerous, benign or undetermined)
2. 18 years of age or older
3. Have been consented to their standard-of-care surgery for resection of the thyroid (partial or complete) and lymph nodes (if applicable)
4. Have had pre-surgical US imaging of the thyroid and lymph nodes

Exclusion Criteria:

1. Inability to provide informed consent
2. Pre-operative therapy for current thyroid cancer (including chemotherapy, endocrine therapy and radiotherapy)
3. History of photosensitivity or skin disease (exposure to laser light is involved in PA imaging)
4. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Detect/localize thyroid nodules and lymph nodes in vivo by using tri-modal imaging | up to 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada